CLINICAL TRIAL: NCT04522973
Title: The Impact of Oral Ethanol and Vaped Ethanol on the Evaluation of Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: U.S. Department of Justice (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HM20018402; 2019-MU-MU-0007 (Other Grant/Funding Number: Department of Justice)
Record Dates: First submitted 2020-08-13; First posted 2020-08-21 (Actual); Results first posted 2025-11-05 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Electronic Cigarette Use
MeSH Terms: conditions — Vaping | interventions — Beverages; Ethanol

STUDY DESIGN:
Intervention Model Description: Single group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Within group four condition comparison (Other): Participants completed four ~5-hour, Latin-square ordered sessions separated by ≥48 hours. Session order was not recorded as it was not relevant to the study outcomes: Beverage with ethanol and E-cigarette liquid with ethanol, Beverage with ethanol and E-cigarette liquid without ethanol, Beverage without ethanol and E-cigarette liquid with ethanol, and Beverage without ethanol and E-cigarette liquid without ethanol.
  Interventions: Other: Beverage with ethanol and E-cigarette liquid with ethanol; Other: Beverage with ethanol and E-cigarette liquid without ethanol; Other: Beverage without ethanol and E-cigarette liquid with ethanol; Other: Beverage without ethanol and E-cigarette liquid without ethanol

INTERVENTIONS:
Other: Beverage with ethanol and E-cigarette liquid with ethanol — Beverage with ethanol and E-cigarette liquid with ethanol
Other: Beverage with ethanol and E-cigarette liquid without ethanol — Beverage with ethanol and E-cigarette liquid without ethanol
Other: Beverage without ethanol and E-cigarette liquid with ethanol — Beverage without ethanol and E-cigarette liquid with ethanol
Other: Beverage without ethanol and E-cigarette liquid without ethanol — Beverage without ethanol and E-cigarette liquid without ethanol

SUMMARY:
The purpose of this research study is to determine if ethanol-containing e-cigarettes impact ethanol breath, blood or oral fluid tests, field sobriety tests, or other tests of sobriety. Ethanol is a common part of e-cigarette liquids.

ELIGIBILITY:
Inclusion Criteria:

* e-cigarette users
* alcohol consumers
* willing to provide informed consent
* able to attend the lab sessions as needed
* agree to use designated products according to study protocol.

Exclusion Criteria:

- Women who are breast-feeding or test positive for pregnancy (by urinalysis) at screening.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Breland, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Within Group Four Condition Comparison: Participants completed four ~5-hour, Latin-square ordered sessions separated by ≥48 hours. Session order was not recorded as it was not relevant to the study outcomes. Session interventions were as follows:
  * Placebo drink: Placebo vape (Beverage without ethanol and E-cigarette liquid without ethanol)
  * Placebo drink: Active vape (Beverage without ethanol and E-cigarette liquid with 20% ethanol)
  * Active drink: Placebo vape (Beverage with 50% ethanol (dosed to have the participant reach a 0.08% BAC) and E-cigarette liquid without ethanol)
  * Active drink: Active vape (Beverage with 50% ethanol (dosed to have the participant reach a 0.08% BAC) and E-cigarette liquid with 20% ethanol)
Period: Overall Study
Arm/Group | Within Group Four Condition Comparison
Started | 12
Completed | 7
Not Completed | 5
Not completed — Lost to Follow-up | 4
Not completed — Could not adhere to study schedule | 1

BASELINE CHARACTERISTICS:
Arm/Group | Within Group Four Condition Comparison
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.6 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Blood Alcohol Concentration
Description: Blood alcohol concentration (BAC) level was determined 6 times over 6 hours to assess for changes in BAC from use of an e-cigarette containing ethanol compared to the use of an e-cigarette without ethanol.
Time Frame: Blood collected before (baseline) and after (0, 40, 55, 200, 215) drinking. The e-cigarette was used at 50 and 210 minutes post-drinking.
Population: Blood Alcohol Concentration (% alcohol)
Measure: Mean (Standard Deviation); unit: percent alcohol
Groups:
- Placebo Drink: Placebo Vape: Beverage without ethanol and E-cigarette liquid without ethanol
- Placebo Drink: Active Vape: Beverage without ethanol and E-cigarette liquid with 20% ethanol
- Active Drink: Placebo Vape: Beverage with 50% ethanol (dosed to have the participant reach a 0.08% BAC) and E-cigarette liquid without ethanol
- Active Drink: Active Vape: Beverage with 50% ethanol (dosed to have the participant reach a 0.08% BAC) and E-cigarette liquid with 20% ethanol
Arm/Group | Placebo Drink: Placebo Vape | Placebo Drink: Active Vape | Active Drink: Placebo Vape | Active Drink: Active Vape
Number analyzed (Participants) | 7 | 7 | 7 | 7
percent alcohol
  Baseline Collection | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  0 Minute Collection Post-Drinking | 0 (0) | 0 (0) | .070 (.037) | .061 (.045)
  40 Minute Collection Post-Drinking | 0 (0) | 0 (0) | .080 (.022) | .088 (.045)
  55 Minute Collection Post-Drinking | 0 (0) | 0 (0) | .072 (.016) | .075 (.008)
  200 Minute Collection Post-Drinking | 0 (0) | 0 (0) | .037 (.013) | .039 (.009)
  210 Minute Collection Post-Drinking | 0 (0) | 0 (0) | .032 (.013) | .034 (.011)

2. Primary Outcome: Breath Alcohol Concentration
Description: Breath Alcohol Concentration (BrAC) was assessed 12 times over 6 hours to determine changes in BrAC from the use of an e-cigarette containing ethanol compared to the use of an e-cigarette without ethanol.
Time Frame: Breath was analyzed before (baseline) and after (10, 20, 40, 55, 90, 120, 165, 200, 215, 240, 270 min) drinking. The e-cigarette was used by the participants at 50 and 210 minutes post-drinking.
Population: Blood Alcohol Concentration (% alcohol)
Measure: Mean (Standard Deviation); unit: percent alcohol
Arm/Group | Placebo Drink: Placebo Vape | Placebo Drink: Active Vape | Active Drink: Placebo Vape | Active Drink: Active Vape
Number analyzed (Participants) | 7 | 7 | 7 | 7
percent alcohol
  Baseline | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  10 minute collection post-drinking | 0 (0) | 0 (0) | .069 (.024) | .080 (.0245)
  20 minute collection post-drinking | 0 (0) | 0 (0) | .071 (.024) | .079 (.025)
  40 minute collection post-drinking | 0 (0) | 0 (0) | .067 (.014) | .073 (.012)
  55 minute collection post-drinking | 0 (0) | 0 (0) | .054 (.012) | .061 (.005)
  90 minute collection post-drinking | 0 (0) | 0 (0) | .049 (.011) | .053 (.008)
  120 minute collection post-drinking | 0 (0) | 0 (0) | .042 (.010) | .045 (.009)
  165 minute collection post-drinking | 0 (0) | 0 (0) | .033 (.009) | .035 (.007)
  200 minute collection post-drinking | 0 (0) | 0 (0) | .026 (.009) | .027 (.008)
  215 minute collection post-drinking | 0 (0) | 0 (0) | .018 (.006) | .024 (.005)
  240 minute collection post-drinking | 0 (0) | 0 (0) | .016 (.010) | .016 (011)
  270 minute collection post-drinking | 0 (0) | 0 (0) | .009 (.009) | .011 (.009)

3. Primary Outcome: Oral Fluid Alcohol Concentration (OFAC)
Description: Oral fluid alcohol concentration (OFAC) was assessed 9 times over 6 hours to determine changes in OFAC from the use of an e-cigarette containing ethanol compared to use of an e-cigarette without ethanol.
Time Frame: Oral fluid was collected before (baseline) and after (0, 5, 20, 40, 55, 200, 215, 240 min) drinking. The e-cigarette was used by the participants at 50 and 210 minutes post-drinking.
Population: Blood Alcohol Concentration (% alcohol)
Measure: Mean (Standard Deviation); unit: Percent Alcohol
Arm/Group | Placebo Drink: Placebo Vape | Placebo Drink: Active Vape | Active Drink: Placebo Vape | Active Drink: Active Vape
Number analyzed (Participants) | 7 | 7 | 7 | 7
Percent Alcohol
  Baseline Collection | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  0 minute collection post-drinking | 0 (0) | 0 (0) | .146 (.075) | .124 (.025)
  5 minute collection post-drinking | 0 (0) | 0 (0) | .118 (.055) | .106 (.052)
  20 minute collection post-drinking | 0 (0) | 0 (0) | .102 (.043) | .109 (.021)
  40 minute collection post-drinking | 0 (0) | 0 (0) | .092 (.031) | .104 (.018)
  55 minute collection post-drinking | 0 (0) | 0 (0) | .081 (.025) | .091 (.017)
  200 minute collection post-drinking | 0 (0) | 0 (0) | .036 (.014) | .040 (.013)
  215 minute collection post-drinking | 0 (0) | 0 (0) | .032 (.020) | .033 (.019)
  240 minute collection post-drinking | 0 (0) | 0 (0) | .023 (.019) | .023 (.018)

4. Primary Outcome: Ethanol Biomarker (5-Hydroxytryptophol) in Blood
Description: 5-Hydroxytryptophol was analyzed in blood 6 times over a course of 6 hours to assess changes in determined concentrations from use of an electronic cigarette containing ethanol.
Time Frame: Blood was collected before (baseline) and after (0, 40, 55, 200, 215 min) drinking. The e-cigarette was used by the participants at 50 and 210 minutes post-drinking.
Population: Ethanol Biomarker (5-Hydroxytryptophol) ng/mL
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Active Drink: Active Vape: dosed to have the participant reach a 0.08% BAC) and E-cigarette liquid with 20% ethanol
Arm/Group | Placebo Drink: Placebo Vape | Placebo Drink: Active Vape | Active Drink: Placebo Vape | Active Drink: Active Vape
Number analyzed (Participants) | 7 | 7 | 7 | 7
ng/mL
  Baseline Collection | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  0 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  40 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  55 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  200 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  215 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)

5. Primary Outcome: Ethanol Biomarkers (5-Hydroxyindoleacetic Acid) in Blood
Description: 5-Hydroxyindoleacetic acid was analyzed in blood 6 times over a course of 6 hours to assess changes in determined concentrations from use of an electronic cigarette containing ethanol.
Time Frame: as for outcome 4
Population: Ethanol Biomarkers (5-Hydroxyindoleacetic Acid) ng/mL
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo Drink: Placebo Vape | Placebo Drink: Active Vape | Active Drink: Placebo Vape | Active Drink: Active Vape
Number analyzed (Participants) | 7 | 7 | 7 | 7
ng/mL
  Baseline Collection | 80 (81) | 90 (91) | 44 (75) | 121 (149)
  0 minute collection post-drinking | 91 (97) | 34 (59) | 44 (29) | 76 (36)
  40 minute collection post-drinking | 97 (96) | 93 (93) | 30 (51) | 63 (81)
  55 minute collection post-drinking | 103 (103) | 75 (99) | 61 (80) | 0 (0)
  200 minute collection post-drinking | 123 (98) | 132 (103) | 71 (94) | 90 (86)
  215 minute collection post-drinking | 82 (81) | 106 (79) | 73 (97) | 83 (114)

6. Primary Outcome: Ethanol Biomarkers (Ethyl Sulfate) Analyzed in Blood/ E-cig Containing Ethanol
Description: Ethyl sulfate was analyzed in blood 6 times over a course of 6 hours to assess changes in determined concentrations from use of an electronic cigarette containing ethanol.
Time Frame: as for outcome 4
Population: Ethanol Biomarkers (Ethyl Sulfate) ng/mL
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo Drink: Placebo Vape | Placebo Drink: Active Vape | Active Drink: Placebo Vape | Active Drink: Active Vape
Number analyzed (Participants) | 7 | 7 | 7 | 7
ng/mL
  Baseline Collection | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  0 minute collection post-drinking | 0 (0) | 0 (0) | 16 (28) | 10 (26)
  40 minute collection post-drinking | 0 (0) | 0 (0) | 167 (80) | 184 (52)
  55 minute collection post-drinking | 0 (0) | 0 (0) | 207 (67) | 211 (46)
  200 minute collection post-drinking | 0 (0) | 0 (0) | 228 (68) | 239 (55)
  215 minute collection post-drinking | 0 (0) | 0 (0) | 218 (67) | 224 (50)

7. Primary Outcome: Ethanol Biomarkers (Phosphatidylethanol 16:0-18:1) in Blood
Description: Phosphatidylethanol 16:0-18:1 was analyzed in blood 6 times over a course of 6 hours to assess changes in determined concentrations from use of an electronic cigarette containing ethanol.
Time Frame: as for outcome 4
Population: Ethanol Biomarkers (Phosphatidylethanol 16:0-18:1) in Blood ng/mL
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo Drink: Placebo Vape | Placebo Drink: Active Vape | Active Drink: Placebo Vape | Active Drink: Active Vape
Number analyzed (Participants) | 7 | 7 | 7 | 7
ng/mL
  Baseline Collection | 402 (438) | 416 (432) | 647 (790) | 409 (323)
  0 minute collection post-drinking | 338 (443) | 304 (433) | 487 (570) | 318 (269)
  40 minute collection post-drinking | 345 (460) | 322 (442) | 562 (688) | 306 (270)
  55 minute collection post-drinking | 330 (401) | 292 (339) | 589 (699) | 374 (284)
  200 minute collection post-drinking | 352 (489) | 302 (353) | 547 (722) | 319 (297)
  215 minute collection post-drinking | 639 (739) | 411 (397) | 718 (744) | 450 (239)

8. Primary Outcome: Ethanol Biomarkers (Phosphatidylethanol 16:0-18:2) in Blood
Description: Phosphatidylethanol 16:0-18:2 was analyzed in blood 6 times over a course of 6 hours to assess changes in determined concentrations from use of an electronic cigarette containing ethanol.
Time Frame: as for outcome 4
Population: Ethanol Biomarkers (Phosphatidylethanol 16:0-18:2) in Blood ng/mL
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo Drink: Placebo Vape | Placebo Drink: Active Vape | Active Drink: Placebo Vape | Active Drink: Active Vape
Number analyzed (Participants) | 7 | 7 | 7 | 7
ng/mL
  Baseline Collection | 894 (956) | 1013 (1403) | 1256 (1756) | 938 (784)
  0 minute collection post-drinking | 549 (757) | 549 (894) | 771 (939) | 616 (577)
  40 minute collection post-drinking | 563 (806) | 572 (768) | 927 (1214) | 617 (589)
  55 minute collection post-drinking | 574 (758) | 466 (580) | 862 (1061) | 832 (587)
  200 minute collection post-drinking | 636 (1000) | 494 (685) | 1028 (1479) | 602 (500)
  215 minute collection post-drinking | 1630 (2090) | 889 (873) | 1544 (1417) | 1081 (480)

9. Primary Outcome: Ethanol Biomarkers (5-Hydroxytryptophol Glucuronide) Analyzed in Blood
Description: 5-Hydroxytryptophol glucuronide was analyzed in blood 6 times over a course of 6 hours to assess changes in determined concentrations from use of an electronic cigarette containing ethanol.
Time Frame: Blood collected before (baseline) and after (0, 40, 55, 200, 215 min) drinking. The e-cigarette was used by the participants at 50 and 210 minutes post-drinking.
Population: Ethanol Biomarkers (5-Hydroxytryptophol Glucuronide) in Blood ng/mL
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo Drink: Placebo Vape | Placebo Drink: Active Vape | Active Drink: Placebo Vape | Active Drink: Active Vape
Number analyzed (Participants) | 7 | 7 | 7 | 7
ng/mL
  Baseline collection | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  0 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  40 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  55 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  200 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  215 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)

10. Primary Outcome: Ethanol Biomarkers (5-Hydroxytryptophol) in Blood
Description: Ethyl glucuronide was analyzed in blood 6 times over a course of 6 hours to assess changes in determined concentrations from use of an electronic cigarette containing ethanol.
Time Frame: as for outcome 9
Population: Ethanol Biomarkers (Ethyl Glucuronide ) in Blood ng/mL
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo Drink: Placebo Vape | Placebo Drink: Active Vape | Active Drink: Placebo Vape | Active Drink: Active Vape
Number analyzed (Participants) | 7 | 7 | 7 | 7
ng/mL
  Baseline | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  0 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  40 minute collection post-drinking | 0 (0) | 0 (0) | 145 (53) | 128 (29)
  55 minute collection post-drinking | 0 (0) | 0 (0) | 175 (52) | 187 (41)
  200 minute collection post-drinking | 0 (0) | 0 (0) | 331 (88) | 406 (104)
  215 minute collection post-drinking | 0 (0) | 0 (0) | 325 (94) | 337 (116)

11. Primary Outcome: Ethanol Biomarkers (5-Hydroxytryptophol) in Analyzed in Oral Fluid
Description: 5-Hydroxyindoleacetic acid was analyzed in oral fluid 9 times over a course of 6 hours to assess changes in determined concentrations from use of an electronic cigarette containing ethanol.
Time Frame: as for outcome 3
Population: Ethanol Biomarkers (5-Hydroxytryptophol) in Oral Fluid ng/mL
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo Drink: Placebo Vape | Placebo Drink: Active Vape | Active Drink: Placebo Vape | Active Drink: Active Vape
Number analyzed (Participants) | 7 | 7 | 7 | 7
ng/mL
  Baseline | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  0 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  5 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  20 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  40 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  55 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  200 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  215 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  240 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)

12. Primary Outcome: Ethanol Biomarkers (5-Hydroxyindoleacetic Acid) Analyzed in Oral Fluid
Description: as for outcome 11
Time Frame: as for outcome 3
Population: Ethanol Biomarkers (5-Hydroxyindoleacetic Acid) in Oral Fluid ng/mL
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo Drink: Placebo Vape | Placebo Drink: Active Vape | Active Drink: Placebo Vape | Active Drink: Active Vape
Number analyzed (Participants) | 7 | 7 | 7 | 7
ng/mL
  Baseline Collection | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  0 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  5 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  20 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  40 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  55 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  200 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  215 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  240 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)

13. Primary Outcome: Ethanol Biomarkers (Ethyl Sulfate) Analyzed in Oral Fluid
Description: Ethyl sulfate was analyzed in oral fluid 9 times over a course of 6 hours to assess changes in determined concentrations from use of an electronic cigarette containing ethanol.
Time Frame: Oral fluid was collected before (baseline) and after (0, 5, 20, 40, 55, 200, 215, 240 min) drinking. The e-cigarette was used by the participant at 50 and 210 minutes post-drinking
Population: Ethanol Biomarkers (Ethyl Sulfate) in Oral Fluid ng/mL
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo Drink: Placebo Vape | Placebo Drink: Active Vape | Active Drink: Placebo Vape | Active Drink: Active Vape
Number analyzed (Participants) | 7 | 7 | 7 | 7
ng/mL
  Baseline Collection | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  0 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  5 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  20 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  40 minute collection post-drinking | 0 (0) | 0 (0) | 8 (21) | 0 (0)
  55 minute collection post-drinking | 0 (0) | 0 (0) | 26 (49) | 8 (21)
  200 minute collection post-drinking | 0 (0) | 0 (0) | 25 (47) | 53 (103)
  215 minute collection post-drinking | 0 (0) | 0 (0) | 29 (37) | 19 (33)
  240 minute collection post-drinking | 0 (0) | 0 (0) | 33 (61) | 44 (58)

14. Primary Outcome: Ethanol Biomarkers (Phosphatidylethanol 16:0-18:1) Analyzed in Blood
Description: Phosphatidylethanol 16:0-18:1 was analyzed in oral fluid 9 times over a course of 6 hours to assess changes in determined concentrations from use of an electronic cigarette containing ethanol.
Time Frame: as for outcome 3
Population: Ethanol Biomarkers (Phosphatidylethanol 16:0-18:1) in Oral Fluid ng/mL
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo Drink: Placebo Vape | Placebo Drink: Active Vape | Active Drink: Placebo Vape | Active Drink: Active Vape
Number analyzed (Participants) | 7 | 7 | 7 | 7
ng/mL
  Baseline Collection | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  0 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  5 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  20 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  40 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  55 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  200 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  215 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  240 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)

15. Primary Outcome: Ethanol Biomarkers (Phosphatidylethanol 16:0-18:2) in Oral Fluid
Description: Phosphatidylethanol 16:0-18:2 was analyzed in oral fluid 9 times over a course of 6 hours to assess changes in determined concentrations from use of an electronic cigarette containing ethanol.
Time Frame: as for outcome 3
Population: Ethanol Biomarkers (Phosphatidylethanol 16:0-18:2) in Oral Fluid ng/mL
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo Drink: Placebo Vape | Placebo Drink: Active Vape | Active Drink: Placebo Vape | Active Drink: Active Vape
Number analyzed (Participants) | 7 | 7 | 7 | 7
ng/mL
  Baseline Collection | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  0 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  20 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  40 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  55 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  200 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  215 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  240 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)

16. Primary Outcome: Ethanol Biomarkers (Ethyl Glucuronide) Analyzed in Blood
Description: as for outcome 10
Time Frame: Blood collected before (baseline) and after (0, 40, 55, 200, 215 min) drinking. The e-cigarette was used by the participant at 50 and 210 minutes post-drinking.
Population: Ethanol Biomarkers (5-Hydroxytryptophol Glucuronide) ng/mL
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Placebo Drink: Placebo Vape: On four separate occasions, participants will come to the research center and complete one of the four conditions. All participants will complete all four study conditions. Sessions will be ordered by Latin-square. Participants will not be assigned to arms based on session order and session order will not be recorded as it is not relevant to the study outcomes.
  Beverage with ethanol and E-cigarette liquid with ethanol: Beverage with ethanol and E-cigarette liquid with ethanol
  Beverage with ethanol and E-cigarette liquid without ethanol: Beverage with ethanol and E-cigarette liquid without ethanol
  Beverage without ethanol and E-cigarette liquid with ethanol: Beverage without ethanol and E-cigarette liquid with ethanol
  Beverage without ethanol and E-cigarette liquid without ethanol: Beverage without ethanol and E-cigarette liquid without ethanol
- Placebo Drink: Active Vape; Active Drink: Placebo Vape; Active Drink: Active Vape: On four separate occasions, participants will come to the research center and complete one of the four conditions. All participants will complete all four study conditions. Sessions will be ordered by Latin-square. Participants will not be assigned to arms based on session order and session order will not be recorded as it is not relevant to the study outcomes.
Arm/Group | Placebo Drink: Placebo Vape | Placebo Drink: Active Vape | Active Drink: Placebo Vape | Active Drink: Active Vape
Number analyzed (Participants) | 7 | 7 | 7 | 7
ng/mL
  Baseline Collection | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  0 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  5 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  20 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  40 minute collection post-drinking | 0 (0) | 0 (0) | 145 (53) | 128 (29)
  55 minute collection post-drinking | 0 (0) | 0 (0) | 175 (52) | 187 (41)
  200 minute collection post-drinking | 0 (0) | 0 (0) | 331 (88) | 406 (104)
  215 minute collection post-drinking | 0 (0) | 0 (0) | 325 (94) | 337 (116)
  240 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)

17. Primary Outcome: Ethanol Biomarkers (Ethyl Glucuronide) Analyzed in Oral Fluid
Description: Ethyl glucuronide was analyzed in oral fluid 9 times over a course of 6 hours to assess changes in determined concentrations from use of an electronic cigarette containing ethanol.
Time Frame: as for outcome 13
Population: Ethanol Biomarkers (Ethyl Glucuronide) in Oral Fluid ng/mL
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo Drink: Placebo Vape | Placebo Drink: Active Vape | Active Drink: Placebo Vape | Active Drink: Active Vape
Number analyzed (Participants) | 7 | 7 | 7 | 7
ng/mL
  Baseline Collection | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  0 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  5 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  20 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  40 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  55 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  200 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  215 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  240 minute collection post-drinking | 0 (0) | 0 (0) | 0 (0) | 0 (0)

18. Secondary Outcome: Horizontal Gaze Nystagmus
Description: Standard Field Sobriety Tests (SFSTs) were administered 4 times over a course of 6 hours to assess changes in objective impairment. The SFST includes the Horizontal Gaze Nystagmus (a jerking or stuttering type of movement observed in a person's eyes that occurs as a result of consuming alcohol or other nervous system depressants) test. For each test, a law enforcement officer records the number of clues observed. HGN has a maximum of 6 clues, 3 per eye:
  1. lack of smooth pursuit
  2. distinct and sustained nystagmus at maximum deviation
  3. onset of nystagmus prior to 45 degrees.
Time Frame: Conducted before drinking (baseline), at 20 minutes post-drinking (before first vaping bout), at 55 minutes post-drinking (after the first vaping), and at 215 minutes post-drinking (after second vaping bout).
Population: Horizontal Gaze Nystagmus # of clues observed
Measure: Mean (Standard Deviation); unit: Number of Clues Observed
Arm/Group | Placebo Drink: Placebo Vape | Placebo Drink: Active Vape | Active Drink: Placebo Vape | Active Drink: Active Vape
Number analyzed (Participants) | 7 | 7 | 7 | 7
Number of Clues Observed
  Baseline | 0 (0) | .9 (.9) | .7 (1.0) | .3 (.8)
  Before the 1st Vaping Bout | .4 (.8) | .9 (.9) | 3.1 (2.1) | 3.9 (1.7)
  After the 1st Vaping Bout | .4 (.8) | .9 (1.1) | 3.0 (1.8) | 3.4 (1.7)
  After the 2nd Vaping Bout | .3 (.8) | 1.1 (1.5) | .7 (1.0) | 1.9 (1.3)

19. Secondary Outcome: Walk and Turn Test
Description: Standard Field Sobriety Tests (SFSTs) were administered 4 times over a course of 6 hours to assess changes in objective impairment. The SFST includes the walk and turn test (suspect to perform a physical task while simultaneously following instructions and maintaining balance; involves walking a straight line heel-to-toe, turning, and walking back, with officers looking for specific indicators of impairment). For each test, a law enforcement officer records the number of clues observed. WAT has a maximum of 8 clues:
  1. inability to balance during the instruction phase
  2. starting before the officer has finished the instructions
  3. Stopping while walking to regain balance
  4. Not touching heel-to-toe
  5. Stepping off the line
  6. Using arms to balance
  7. Losing balance on the turn or turning incorrectly
  8. Taking the wrong number of steps
Time Frame: as for outcome 18
Population: Walk and Turn Test, # of clues observed
Measure: Mean (Standard Deviation); unit: Number of Clues Observed
Arm/Group | Placebo Drink: Placebo Vape | Placebo Drink: Active Vape | Active Drink: Placebo Vape | Active Drink: Active Vape
Number analyzed (Participants) | 7 | 7 | 7 | 7
Number of Clues Observed
  Baseline | .6 (.8) | .9 (1.1) | .9 (.9) | .6 (.5)
  Before the 1st Vaping Bout | .4 (.8) | .9 (.7) | 1.1 (1.3) | 1.1 (1.2)
  After the 1st Vaping Bout | .3 (.5) | .4 (.8) | 1.0 (1.3) | 1.1 (1.1)
  After the 2nd Vaping Bout | .1 (.4) | .7 (.8) | .6 (.5) | .7 (.8)

20. Secondary Outcome: One Leg Stand Test
Description: Standard Field Sobriety Tests (SFSTs) were administered 4 times over a course of 6 hours to assess changes in objective impairment. The SFST includes the one-leg stand test (assess balance and coordination, potentially indicating impairment due to alcohol or drugs). For each test, a law enforcement officer records the number of clues observed. OLS has a maximum of 4 clues: Swaying while balancing, Using arms for balance, Hopping 4. Putting the raised foot down
Time Frame: as for outcome 18
Population: One leg stand test, # of clues observed
Measure: Mean (Standard Deviation); unit: Number of Clues observed
Arm/Group | Placebo Drink: Placebo Vape | Placebo Drink: Active Vape | Active Drink: Placebo Vape | Active Drink: Active Vape
Number analyzed (Participants) | 7 | 7 | 7 | 7
Number of Clues observed
  Baseline | .6 (.8) | .7 (1.1) | .4 (.5) | .7 (.8)
  Before the 1st Vaping Bout | .3 (.5) | 0 (0) | .9 (1.5) | 1 (1.3)
  After the 1st Vaping Bout | .6 (.8) | .3 (.5) | .4 (.8) | 1.1 (1.3)
  After the 2nd Vaping Bout | .6 (.8) | .3 (.5) | .3 (.5) | .4 (.8)

21. Other Pre Specified Outcome: Subjective High Assessment Scale Questionnaire (SHAS)
Description: Subjective High Assessment Scale Questionnaire (SHAS) is a 14-item questionnaire used to assess how intoxicated a person feels after consuming alcohol, typically administered in laboratory settings. It focuses on capturing subjective sensations associated with intoxication, such as feeling "clumsy," "dizzy," or "high". Participants rate their experience on a visual analog scale (a line with markings) to indicate the extent to which they feel each symptom at a given time. The scale ranges from Normal" (0) to "Extremely" (100). The score for each of the questions is summed to give an overall indication of the individual's subjective intoxication. A higher score would indicate greater feelings of impairment.
Time Frame: Administered at baseline, 55 minutes post-drinking (after first vape bout), and 215 minutes post-drinking (after second vape bout).
Population: Subjective High Assessment Scale Questionnaire (SHAS) Total score
Measure: Mean (Standard Deviation); unit: SHAS Total score
Arm/Group | Placebo Drink: Placebo Vape | Placebo Drink: Active Vape | Active Drink: Placebo Vape | Active Drink: Active Vape
Number analyzed (Participants) | 7 | 7 | 7 | 7
SHAS Total score
  Baseline | 60 (74) | 58 (75) | 38 (41) | 29 (30)
  After e-cig use at 55 minutes | 91 (64) | 78 (71) | 244 (271) | 286 (241)
  After e-cig use at 215 minutes | 52 (47) | 48 (51) | 105 (132) | 172 (229)

22. Other Pre Specified Outcome: Biphasic Alcohol Effects Scale Questionnaire (BAES)
Description: Biphasic Alcohol Effects Scale Questionnaire (BAES) is a 14-item questionnaire consisting of adjectives that describe the stimulant- and sedative-like effects of alcohol. The items are presented in alphabetical order, and are rated on an 11-point rating scale from 0=Not at All to 10=Extremely. The score for each of the questions was summed to give an overall indication of the individual's subjective intoxication. A higher score would indicate greater feelings of impairment.
Time Frame: as for outcome 21
Population: Biphasic Alcohol Effects Scale Questionnaire (BAES) total score
Measure: Mean (Standard Deviation); unit: (BAES) total score
Arm/Group | Placebo Drink: Placebo Vape | Placebo Drink: Active Vape | Active Drink: Placebo Vape | Active Drink: Active Vape
Number analyzed (Participants) | 7 | 7 | 7 | 7
(BAES) total score
  Baseline | 22 (15) | 25 (11) | 28 (15) | 25 (14)
  After e-cig use at 55 minutes | 22 (11) | 25 (11) | 33 (17) | 36 (14)
  After e-cig use at 215 minutes | 24 (14) | 24 (14) | 28 (12) | 32 (12)

23. Other Pre Specified Outcome: General Labeled Magnitude Scale Questionnaire (gLMS)
Description: The general labeled magnitude scale (gLMS) is a psychophysical scaling method used to measure the perceived intensity of various sensations. A gLMS typically ranges from 0 (undetectable) to 100 (strongest imaginable sensation/experience of any kind). Crucially, it uses specific labels positioned at specific points on the scale (e.g., barely detectable, weak, moderate, strong, very strong). The gLMS was comprised of 3 questions asking participants to indicate the overall flavor sensation, harshness, and throat hit of the e-cigarette. The score for each of the questions was summed. A higher score would indicate greater sensations from e-cigarette use.
Time Frame: as for outcome 21
Population: General Labeled Magnitude Scale Questionnaire (gLMS) total score
Measure: Mean (Standard Deviation); unit: (gLMS) total score
Arm/Group | Placebo Drink: Placebo Vape | Placebo Drink: Active Vape | Active Drink: Placebo Vape | Active Drink: Active Vape
Number analyzed (Participants) | 7 | 7 | 7 | 7
(gLMS) total score
  Baseline | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  After e-cig use at 55 minutes | 91 (51) | 108 (58) | 86 (66) | 105 (57)
  After e-cig use at 215 minutes | 83 (63) | 105 (67) | 101 (61) | 81 (69)

24. Other Pre Specified Outcome: Labeled Hedonic Scale Questionnaire (LHS)
Description: A survey tool used to measure how much someone likes or dislikes something using descriptive labels for different levels of liking and disliking. Instead of just numbers, the scale uses words or phrases that describe the intensity of liking or disliking (e.g., "most disliked sensation imaginable"=0, "neutral" = 50, and "most liked sensation imaginable"=100) and aim to provide ratio-level data, meaning that the differences between scale points are meaningful and proportional. the LHS was comprised of 4 questions asking participants to indicate the e-cigarette's overall flavor sensation, harshness, throat hit, and warmth of the vapor. The score for each of the questions was summed. A higher score would indicate a more liked overall vaping experience; a lower score would indicate a more disliked overall vaping experience
Time Frame: as for outcome 21
Population: Labeled Hedonic Scale Questionnaire (LHS) total score
Measure: Mean (Standard Deviation); unit: (LHS) total score
Arm/Group | Placebo Drink: Placebo Vape | Placebo Drink: Active Vape | Active Drink: Placebo Vape | Active Drink: Active Vape
Number analyzed (Participants) | 7 | 7 | 7 | 7
(LHS) total score
  Baseline | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  After e-cig use at 55 minutes | 161 (37) | 125 (42) | 184 (71) | 165 (66)
  After e-cig use at 215 minutes | 180 (44) | 121 (55) | 152 (81) | 152 (61)

25. Other Pre Specified Outcome: Direct Effects of Vaping Questionnaire (DEPVQ)
Description: Direct Effects of Vaping Questionnaire (DEVQ) is a 10-item Questionnaire that asks participants about their vaping experience (10 questions, each scored from 0 - 100). While subscale scores are often the primary focus, an overall score may be calculated by summing all item scores or averaging them. The score for each of the questions was summed. A higher score indicates the e-cigarette evoked greater subjective effects or feelings.
Time Frame: as for outcome 21
Population: Direct Effects of Vaping Questionnaire (DEPVQ) total score
Measure: Mean (Standard Deviation); unit: (DEPVQ) total score
Arm/Group | Placebo Drink: Placebo Vape | Placebo Drink: Active Vape | Active Drink: Placebo Vape | Active Drink: Active Vape
Number analyzed (Participants) | 7 | 7 | 7 | 7
(DEPVQ) total score
  Baseline | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  After e-cig use at 55 minutes | 320 (132) | 259 (151) | 289 (183) | 309 (136)
  After e-cig use at 215 minutes | 255 (117) | 205 (108) | 259 (112) | 243 (128)

ADVERSE EVENTS:
Time Frame: From baseline to session completion, approximately 7 hours for each session. On average, participants completed all 4 sessions within 1 month.
Arm/Group | Within Group Four Condition Comparison
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 2/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Within Group Four Condition Comparison (N=7)
nausea (Injury, poisoning and procedural complications) | 2 (2) — 1 (14.3%) In the placebo drink/active vape group, 1 (14.3%) in the active drink/placebo vape group

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-09-05): https://cdn.clinicaltrials.gov/large-docs/73/NCT04522973/Prot_001.pdf
  • Informed Consent Form (2023-06-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT04522973/ICF_000.pdf